CLINICAL TRIAL: NCT07153471
Title: A Phase 3 Study to Investigate the Efficacy and Safety of Orforglipron Once Daily in Participants Who Have Obesity or Overweight and Osteoarthritis of the Knee: A Multicenter, Randomized, Double-Blind, Parallel-Arm, Placebo-Controlled Trial
Brief Title: A Study of Orforglipron (LY3502970) in Participants With Obesity or Overweight and Osteoarthritis (OA) of the Knee
Acronym: ATTAIN-OA PAIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27633; 2025-522631-34-00 (EU CTIS Number); J2A-MC-GZPT (Other: Eli Lilly and Company); J2A-MC-GZT1 (Other: Eli Lilly and Company); J2A-MC-GZT2 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-09-02; First posted 2025-09-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis
Keywords: Arthritis; Overnutrition; Nutrition Disorder; Joint Diseases; Musculoskeletal Disease; Knee Degeneration; Osteoarthrosis; Obese
MeSH Terms: conditions — Osteoarthritis; Arthritis; Overnutrition; Nutrition Disorders; Joint Diseases; Musculoskeletal Diseases; Obesity | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orforglipron (GZT1) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (GZT1) (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo
- Orforglipron (GZT2) (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (GZT2) (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: (LY3502970)
  Arms: Orforglipron (GZT1); Orforglipron (GZT2)
Drug: Placebo — Administered orally
  Arms: Placebo (GZT1); Placebo (GZT2)

SUMMARY:
The GZPT master protocol will support two independent studies, J2A-MC-GZT1 and J2A-MC-GZT2. Each study will see how well and safely orforglipron works in people with obesity or overweight who have osteoarthritis (OA) of the knee with pain. Participation in the study will last about 74 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of 27 kilograms per square meter (kg/m2) or higher at screening
* Have tried at least once to lose weight through diet but were unsuccessful
* Have osteoarthritis of the knee and at least one of the following conditions:

  * Be over 50 years old
  * Have morning knee stiffness that lasts about 30 minutes
  * Have a crackling or grinding sound or feeling in the knee

Exclusion Criteria:

* Have gained or lost more than 11 pounds within 90 days prior to screening
* Have had a surgery for obesity or plan to have one in the next 18 months
* Have an active knee infection
* Have type 1 diabetes, type 2 diabetes, or any other type of diabetes
* Have had a recent heart condition or New York Heart Association Functional Classification Class IV congestive heart failure
* Have used any glucagon-like peptide-1 (GLP-1) receptor agonist medication within 180 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score | Baseline, Week 72

SECONDARY OUTCOMES:
Change from Baseline in the WOMAC Physical Function Subscale Score | Baseline, Week 72
Percent Change from Baseline in Body Weight | Baseline, Week 72
Change from Baseline in 36-item, Short-Form Health Survey, version 2 (SF-36v2) Acute Form Physical Functioning Domain Score | Baseline, Week 72
Change from Baseline in Distance Walked During the 6-Minute Walk Test | Baseline, Week 72
Percent Change from Baseline in High-Sensitivity, C-reactive Protein (hsCRP) | Baseline, Week 72
Change from Baseline in Waist Circumference | Baseline, Week 72
Percent Change from Baseline in Tumor Necrosis Factor (TNF)-Alpha | Baseline, Week 72
Change from Baseline in WOMAC Stiffness Subscale | Baseline, Week 72
Change from Baseline in WOMAC Total Score | Baseline, Week 72
Change from Baseline in SF-36v2 Acute Form Domain Scores | Baseline, Week 72
  With exception of the Physical Functioning Domain Score
Percentage of Participants Who Achieve Improved Categorical Shift in Patient Global Impression of Severity (PGIS) - Target Knee Function | Baseline, Week 72
Percentage of Participants Who Achieve Improved Categorical Shift in PGIS - Target Knee Pain | Baseline, Week 72
Change from Baseline in Average Pain Intensity Numeric Rating Scale (API-NRS) Score | Baseline, Week 72
Change from Baseline in Worst Pain Intensity Numeric Rating Scale (WPI-NRS) Score | Baseline, Week 72
Number of Participants with Allowed Concomitant Pain Medication | Baseline, Week 72
Percent Change from Baseline in Total Cholesterol | Baseline, Week 72
Pharmacokinetics (PK): Steady-State Area Under the Curve (AUC) of Orforglipron | Predose through Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (92):
- United States (26):
  - Arizona Research Center, Phoenix, Arizona
  - AMR Clinical, Tempe, Arizona
  - Care Access - Huntington Beach, Huntington Beach, California
  - Care Access - Thousand Oaks, Thousand Oaks, California
  - Legacy Clinical Trials, Colorado Springs, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Care Access - Decatur, Decatur, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Northwestern University, Chicago, Illinois
  - AMR Clinical, Newton, Kansas
  - MedVadis Research Corporation, Waltham, Massachusetts
  - StudyMetrix Research, City of Saint Peters, Missouri
  - AMR Clinical, Kansas City, Missouri
  - Cardio Metabolic Institute, Somerset, New Jersey
  - Carolina Research Center, Shelby, North Carolina
  - University Orthopedics Center, Altoona, Pennsylvania
  - Care Access - Rapid City, Rapid City, South Dakota
  - AMR Clinical, Knoxville, Tennessee
  - Mercy Family Clinic, Dallas, Texas
  - Juno Research, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Activian Clinical Research, Kingwood, Texas
  - Advanced Rheumatology of Houston - Woodlands, The Woodlands, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Gershon Pain Specialists, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (9):
  - Aggarwal and Associates Limited, Brampton
  - Diex Recherche Inc. Division Joliette, Joliette
  - Your Research Network, Niagara Falls
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec
  - Alpha Recherche Clinique, Québec
  - ALPHA Recherche Clinique, Québec
  - Bluewater Clinical Research Group Inc., Sarnia
  - Winterberry Research Inc., Stoney Creek
  - Dr. M.B. Jones Inc., Victoria
- China (12):
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technolo -T, Baotou
  - Xuanwu Hospital Capital Medical University, Beijing
  - The Second Affiliated Hospital Chongqing Medical University, Chongqing
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - The Second People's Hospital of Hefei, Hefei
  - Jinan Central Hospital, Jinan
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - Jiangsu Province Hospital, Nanjing
  - Pingxiang People's Hospital, Pingxiang
  - Huashan Hospital, Fudan University, Shanghai
  - The First Affiliated Hospital of Shantou University Medical College, Shantou
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
- Germany (14):
  - Klinische Forschung Berlin-Mitte, Berlin
  - Siteworks GmbH - Bochum, Bochum
  - Klinische Forschung Dresden, Dresden
  - HRF II - Hamburger Rheuma Forschungszentrum II MVZ für Rheumatologie und Autoimmunmedizin Hamburg GmbH / -T, Hamburg
  - Klinische Forschung Hamburg, Hamburg
  - Klinische Forschung Hannover-Mitte, Hanover
  - Siteworks GmbH - Hannover, Hanover
  - Siteworks GmbH - Heidelberg, Heidelberg
  - Klinische Forschung Karlsruhe, Karlsruhe
  - AmBeNet GmbH, Leipzig
  - CDG Studienambulanz Hartard, München
  - Dedicated Research Site FutureMeds, Offenbach
  - Private Practice - Dr. Jochen Walter, Rendsburg
  - Universitaetsklinikum Wuerzburg, Würzburg
- India (6):
  - All India Institute of Medical Sciences, Bhubaneswar
  - Rajiv Gandhi Government General Hospital, Chennai
  - Atmaram Child Care, Kanpur
  - Kims Kingsway Hospital, Nagpur
  - Maulana Azad Medical College and Associated with Lok Nayak Hospital, New Delhi
  - Vencer Hospital, Pimpri-Chinchwad
- Japan (11):
  - Hamanomachi Hospital, Fukuoka
  - Fukuoka Wajiro Hospital, Fukuoka
  - Shimane University Hospital, Izumo
  - Kariya Toyota General Hospital, Kariya
  - Ando Orthopedic, Kawasaki
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Goto Orthopedic Surgery Clinic, Miyazaki
  - Kato Orthopedic Clinic, Morioka
  - Japan Community Health Care Organization - Saitama Medical Center, Saitama
  - Sapporo Maruyama Orthopedic Hospital, Sapporo
  - Masumoto Orthopedics Clinic, Suginami City
- Mexico (6):
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C., Ciudad Madero
  - Centro Medico del Angel, Mexicali
  - Kohler & Milstein Research S.A. De C.V., Mérida
  - IMED Internal Medicine Clin Trials, Monterrey
  - Clínica García Flores SC, Monterrey
- Spain (8):
  - Hospital San Rafael - La Coruña, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Quirón Málaga, Málaga
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Clínica Gaias - Santiago, Santiago de Compostela
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Quiron Infanta Luisa, Seville
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Orforglipron (LY3502970) in Participants With Obesity or Overweight and Osteoarthritis (OA) of the Knee ( ATTAIN-OA PAIN ) — https://trials.lilly.com/en-US/trial/648295